CLINICAL TRIAL: NCT04560816
Title: A Randomized, 3-Treatment, 3-Period, 6-Sequence, Crossover, Placebo- and Active-Controlled, Double-Blind for ALXN1840 (Open-Label for Moxifloxacin) Thorough QT/QTc Study to Evaluate ALXN1840 on Cardiac Repolarization in Healthy Adults
Brief Title: A Study of the Cardiac Effects of ALXN1840 in Healthy Adults
Status: Completed | Phase: Phase 1 | Type: Interventional
Sponsor: Alexion Pharmaceuticals, Inc. (Industry)
Collaborators: PPD Development, LP (Industry); ERT: Clinical Trial Technology Solutions (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Crossover | Masking: Double | Purpose: Treatment
Other Study IDs: ALXN1840-HV-107
Record Dates: First submitted 2020-09-18; First posted 2020-09-23 (Actual); Results first posted 2023-08-14 (Actual); Last update posted 2023-08-14 (Actual); Status verified 2022-09

CONDITIONS: Healthy
Keywords: Electrocardiogram; Cardiac Repolarization; ALXN1840; Optimized QT Correction; QT Interval Correction; Thorough QT; QT Correction by Fridericia; Individual QT Correction; Wilson Disease
MeSH Terms: conditions — Hepatolenticular Degeneration | interventions — tetrathiomolybdate; Moxifloxacin

STUDY DESIGN:
Intervention Model Description: This will be a 3-treatment, 3-period, 6-sequence, crossover study in healthy adults.
Who Masked: Participant, Care Provider
Masking Description: This study will employ a double-blind study design. The ALXN1840 and matching placebo will be identical in appearance and will be administered in a double-blind manner.
  Moxifloxacin will not be blinded.
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: Yes | FDA-regulated Device: No

ARMS (6):
- Treatment Sequence 1 (Experimental): On Day 1 of each period, participants will receive a single dose of the following study interventions:
  Period 1: ALXN1840.
  Period 2: Placebo-matching ALXN1840.
  Period 3: Moxifloxacin.
  Interventions: Drug: ALXN1840; Drug: Placebo; Drug: Moxifloxacin
- Treatment Sequence 2 (Experimental): On Day 1 of each period, participants will receive a single dose of the following study interventions:
  Period 1: ALXN1840.
  Period 2: Moxifloxacin.
  Period 3: Placebo-matching ALXN1840.
  Interventions: Drug: ALXN1840; Drug: Placebo; Drug: Moxifloxacin
- Treatment Sequence 3 (Experimental): On Day 1 of each period, participants will receive a single dose of the following study interventions:
  Period 1: Placebo-matching ALXN1840.
  Period 2: ALXN1840.
  Period 3: Moxifloxacin.
  Interventions: Drug: ALXN1840; Drug: Placebo; Drug: Moxifloxacin
- Treatment Sequence 4 (Experimental): On Day 1 of each period, participants will receive a single dose of the following study interventions:
  Period 1: Placebo-matching ALXN1840.
  Period 2: Moxifloxacin.
  Period 3: ALXN1840.
  Interventions: Drug: ALXN1840; Drug: Placebo; Drug: Moxifloxacin
- Treatment Sequence 5 (Experimental): On Day 1 of each period, participants will receive a single dose of the following study interventions:
  Period 1: Moxifloxacin.
  Period 2: ALXN1840.
  Period 3: Placebo-matching ALXN1840.
  Interventions: Drug: ALXN1840; Drug: Placebo; Drug: Moxifloxacin
- Treatment Sequence 6 (Experimental): On Day 1 of each period, participants will receive a single dose of the following study interventions:
  Period 1: Moxifloxacin.
  Period 2: Placebo-matching ALXN1840.
  Period 3: ALXN1840.
  Interventions: Drug: ALXN1840; Drug: Placebo; Drug: Moxifloxacin

INTERVENTIONS:
Drug: ALXN1840 — ALXN1840 (120 milligrams) will be administered orally (supratherapeutic dose).
  Other Names: WTX101; Bis-choline tetrathiomolybdate; Tiomolibdate choline
Drug: Placebo — Placebo will be administered orally.
  Other Names: Placebo-matching ALXN1840
Drug: Moxifloxacin — Moxifloxacin (400 milligrams) will be administered orally.

SUMMARY:
This study will evaluate the effect of a supratherapeutic dose of ALXN1840 on the heart rate (HR)-corrected QT interval (QTc) in healthy adult participants. Moxifloxacin will be used as the active control.

DETAILED DESCRIPTION:
This is a randomized, 3-treatment, 3-period, 6-sequence, crossover, placebo- and active-controlled, double-blind for ALXN1840, open-label for moxifloxacin, in healthy adult participants. Participants will be domiciled in the clinic for 7 days during Treatment Period 1 and for 6 days during Treatment Period 2 and 3. A single oral dose of each treatment (ALXN1840, matching ALXN1840 placebo, or moxifloxacin) will be administered on Day 1 of each period following an overnight fast of at least 10 hours. There will be a minimum 14-day washout between study intervention administrations for each treatment period. Cardiodynamic, pharmacokinetic, and safety assessments will be performed at certain times during the study. An end-of-study visit will occur 14 days (±2 days) after the last dose.

ELIGIBILITY:
Inclusion Criteria:

1. Nonsmoker.
2. Body weight at least 60 kilograms (kg) for males or 52 kg for females and body mass index ≥18.0 and ≤30.0 kg/meter squared.
3. Willing and able to follow protocol-specified contraception requirements.
4. Participant has no clinically significant history or presence of ECG findings.

Exclusion Criteria:

1. History or presence of clinical and/or lab disorders.
2. Lymphoma, leukemia, or any malignancy within the past 5 years, or breast cancer within the past 10 years.
3. Participant has abnormal blood pressure, defined as a supine blood pressure <90/50 millimeters of mercury (mm Hg) or >140/90 mm Hg.
4. Serum potassium, calcium, or magnesium levels outside the normal range.
5. Serum copper and/or ceruloplasmin values below the lower limit of normal at Screening.
6. Female participant has hemoglobin <10.8 grams/deciliter (g/dL) and male participant has hemoglobin <12.5 g/dL.
7. Clinically significant multiple or severe allergies.
8. Alanine aminotransferase, aspartate aminotransferase, serum creatinine, or total bilirubin greater than upper limit of normal (with the exception of Gilbert's syndrome).

Ages: 18 Years to 50 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult
Enrollment: 57 (Actual)
Dates: Start 2020-07-24 (Actual); Primary Completion 2021-03-24 (Actual); Study Completion 2021-03-24 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Eugene S. Swenson, MD, PhD, Study Director — Alexion Pharmaceuticals, Inc.; Masood Sadaat, MD, MSc, Study Chair — Alexion Pharmaceuticals, Inc.
Locations (1):
- PPD Development, LP, Austin, Texas, United States

IPD SHARING:
Plan to Share IPD: No

RESULTS

PARTICIPANT FLOW:
Recruitment Details: Only healthy participants were eligible for enrollment. Participants with cardiovascular, respiratory, hepatic, renal, gastrointestinal, endocrine, hematological, psychiatric, or neurologic disorders; abnormal blood pressure, history of cardiac abnormalities, or abnormal clinical laboratory results were excluded from the study.
Pre-assignment Details: One participant was excluded from the pharmacokinetic (PK)/corrected QT interval (QTc) set as a result of having no postdose data for PK concentration and QTc data at matching time points.
Groups:
- Treatment Sequence 1: ABC: On Day 1 of each period, participants received a single dose of the following study interventions:
  Period 1: ALXN1840 120 milligrams (mg) administered as 15 mg enteric-coated tablets (supratherapeutic dose). Period 2: Enteric-coated placebo tablets matching ALXN1840. Period 3: Moxifloxacin 400 mg tablet.
- Treatment Sequence 2: ACB: On Day 1 of each period, participants received a single dose of the following study interventions:
  Period 1: ALXN1840 120 mg administered as 15 mg enteric-coated tablets (supratherapeutic dose). Period 2: Moxifloxacin 400 mg tablet. Period 3: Enteric-coated placebo tablets matching ALXN1840.
- Treatment Sequence 3: BAC: On Day 1 of each period, participants received a single dose of the following study interventions:
  Period 1: Enteric-coated placebo tablets matching ALXN1840. Period 2: ALXN1840 120 mg administered as 15 mg enteric-coated tablets (supratherapeutic dose). Period 3: Moxifloxacin 400 mg tablet.
- Treatment Sequence 4: BCA: On Day 1 of each period, participants received a single dose of the following study interventions:
  Period 1: Enteric-coated placebo tablets matching ALXN1840. Period 2: Moxifloxacin 400 mg tablet. Period 3: ALXN1840 120 mg administered as 15 mg enteric-coated tablets (supratherapeutic dose).
- Treatment Sequence 5: CAB: On Day 1 of each period, participants received a single dose of the following study interventions:
  Period 1: Moxifloxacin 400 mg tablet. Period 2: ALXN1840 120 mg administered as 15 mg enteric-coated tablets (supratherapeutic dose). Period 3: Enteric-coated placebo tablets matching ALXN1840.
- Treatment Sequence 6: CBA: On Day 1 of each period, participants received a single dose of the following study interventions:
  Period 1: Moxifloxacin 400 mg tablet. Period 2: Enteric-coated placebo tablets matching ALXN1840. Period 3: ALXN1840 120 mg administered as 15 mg enteric-coated tablets (supratherapeutic dose).
Period: Overall Study
Arm/Group | Treatment Sequence 1: ABC | Treatment Sequence 2: ACB | Treatment Sequence 3: BAC | Treatment Sequence 4: BCA | Treatment Sequence 5: CAB | Treatment Sequence 6: CBA
Started | 11 | 10 | 8 | 9 | 11 | 8
Completed | 8 | 9 | 7 | 9 | 8 | 8
Not Completed | 3 | 1 | 1 | 0 | 3 | 0
Not completed — Withdrawal by Subject | 1 | 1 | 1 | 0 | 3 | 0
Not completed — Lost to Follow-up | 1 | 0 | 0 | 0 | 0 | 0
Not completed — Protocol Violation | 1 | 0 | 0 | 0 | 0 | 0

BASELINE CHARACTERISTICS:
Population: All participants who received at least 1 dose of ALXN1840 during treatment period.
Groups:
- Overall Study: All participants were randomly assigned to receive a single dose of each the following 3 treatments in 1 of 6 treatment sequences:
  * ALXN1840 120 mg administered as 15 mg enteric-coated tablets (supratherapeutic dose)
  * Enteric-coated placebo tablets matching ALXN1840
  * Moxifloxacin 400 mg tablet
Arm/Group | Overall Study
Number analyzed (Participants) | 57
Age, Continuous [Mean (Standard Deviation); unit: years] | 34.4 (7.63)
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 21
  Male | 36
Ethnicity (NIH/OMB) [Count of Participants; unit: Participants]
  Hispanic or Latino | 22
  Not Hispanic or Latino | 35
  Unknown or Not Reported | 0
Race (NIH/OMB) [Count of Participants; unit: Participants]
  American Indian or Alaska Native | 1
  Asian | 0
  Native Hawaiian or Other Pacific Islander | 0
  Black or African American | 25
  White | 28
  More than one race | 3
  Unknown or Not Reported | 0

OUTCOME MEASURES:

1. Primary Outcome: Placebo-corrected Change From Baseline For QTcF (ΔΔQTcF) for ALXN1840 Using The By-time Point Analysis
Description: Twelve-lead electrocardiograms (ECGs) were extracted from approximately 25-hour continuous (Holter) recordings on Day -1 of Treatment Period 1 and Days 1 and 2 in each treatment period. Change from baseline in the QT interval was corrected for heart rate using Fridericia's formula (ΔQTcF). ΔQTcF was based on a mixed-effects model for repeated measures (MMRM) with ΔQTcF as the dependent variable; period, sequence, time, treatment, and time-by-treatment interaction as fixed effects; and baseline QTc and sex as covariates.
  ΔΔQTc = LS mean ΔQTcF after ALXN1840 dosing minus LS mean ΔQTcF after placebo. If the upper bound of the confidence interval (CI) of ΔΔQTcF was < 10 ms for all postdose time points, ALXN1840 was concluded to not have a significant effect on QT interval prolongation.
Time Frame: Baseline (average of samples taken at -45, -30, and -15 minutes before dosing), 0.5, 1, 2, 3, 4, 5, 6, 7, 8, 10, 12, and 24 (Day 2) hours postdose
Population: All participants who received at least 1 dose of study treatment with measurements at baseline as well as on-treatment with evaluable data at the specified timepoints.
Measure: Least Squares Mean (90% Confidence Interval); unit: ms
Groups:
- ALXN1840: Participants received ALXN1840 120 mg administered as 15 mg enteric-coated tablets (supratherapeutic dose).
Arm/Group | ALXN1840
Number analyzed (Participants) | 57
ms
  Day 1, 0.5 hours postdose | -0.21 [-1.46 to 1.05]
  Day 1, 1 hour postdose | -0.31 [-1.64 to 1.02]
  Day 1, 2 hours postdose | 0.07 [-1.43 to 1.57]
  Day 1, 3 hours postdose | -0.64 [-2.06 to 0.79]
  Day 1, 4 hours postdose | -1.08 [-2.75 to 0.59]
  Day 1, 5 hours postdose | -0.90 [-1.80 to 1.60]
  Day 1, 6 hours postdose | -0.71 [-2.72 to 1.31]
  Day 1, 7 hours postdose | 0.25 [-1.56 to 2.06]
  Day 1, 8 hours postdose | -0.93 [-2.56 to 0.69]
  Day 1, 10 hours postdose | 0.76 [-1.15 to 2.67]
  Day 1, 12 hours postdose | 0.05 [-2.14 to 2.23]
  Day 2, 24 hours postdose | 2.30 [0.85 to 3.74]

2. Secondary Outcome: ΔΔQTcF For Moxifloxacin Using The By-time Point Analysis
Description: Assay sensitivity was evaluated using the by-time point analysis of the effect on ΔΔQTc of moxifloxacin.
  If ΔΔQTcF was larger than 5 ms at 1, 2, and 3 hours postdose, assay sensitivity was considered to be demonstrated.
Time Frame: 1, 2, and 3 hours postdose at Day 1
Population: All participants who received at least 1 dose of moxifloxacin with measurements at baseline as well as on-treatment with evaluable data at the specified timepoints.
Measure: Least Squares Mean (90% Confidence Interval); unit: ms
Groups:
- Moxifloxacin: Participants received moxifloxacin 400 mg tablet.
Arm/Group | Moxifloxacin
Number analyzed (Participants) | 53
ms
  Day 1, 1 hour postdose | 9.65 [8.29 to 11.01]
  Day 1, 2 hours postdose | 11.04 [9.51 to 12.57]
  Day 1, 3 hours postdose | 11.37 [9.91 to 12.83]

3. Secondary Outcome: Change From Baseline For Heart Rate (ΔHR)
Description: Twelve-lead ECGs were extracted from approximately 25-hour continuous (Holter) recordings on Day -1 of Treatment Period 1 and Days 1 and 2 in each treatment period.
Time Frame: Baseline (average of samples taken at 45, -30, and -15 minutes before dosing), 0.5, 1, 2, 3, 4, 5, 6, 7, 8, 10, 12, and 24 (Day 2) hours postdose
Population: as for outcome 1
Measure: Least Squares Mean (90% Confidence Interval); unit: bpm
Groups:
- Placebo: Participants received enteric-coated placebo tablets matching ALXN1840.
Arm/Group | ALXN1840 | Placebo | Moxifloxacin
Number analyzed (Participants) | 57 | 56 | 53
bpm
  Day 1, 0.5 hours postdose | -0.27 [-1.06 to 0.52] | 0.50 [-0.29 to 1.30] | 1.27 [0.45 to 2.09]
  Day 1, 1 hour postdose | -0.02 [-0.90 to 0.85] | 0.38 [-0.50 to 1.26] | 3.87 [2.97 to 4.78]
  Day 1, 2 hours postdose | -0.12 [-0.93 to 0.69] | 0.19 [-0.61 to 1.00] | 1.97 [1.15 to 2.80]
  Day 1, 3 hours postdose | 0.41 [-0.53 to 1.35] | -1.17 [-2.11 to -0.22] | 2.14 [1.17 to 3.12]
  Day 1, 4 hours postdose | 0.51 [-0.50 to 1.52] | 0.24 [-0.77 to 1.25] | 2.30 [1.26 to 3.35]
  Day 1, 5 hours postdose | 5.85 [4.81 to 6.90] | 4.83 [3.78 to 5.87] | 5.82 [4.74 to 6.90]
  Day 1, 6 hours postdose | 7.07 [5.98 to 8.17] | 6.95 [5.86 to 8.03] | 7.43 [6.30 to 8.56]
  Day 1, 7 hours postdose | 5.59 [4.31 to 6.87] | 4.32 [3.03 to 5.61] | 6.61 [5.26 to 7.95]
  Day 1, 8 hours postdose | 4.69 [3.61 to 5.77] | 3.97 [2.89 to 5.05] | 5.37 [4.25 to 6.49]
  Day 1, 10 hours postdose | 7.71 [6.38 to 9.04] | 7.44 [6.09 to 8.79] | 9.15 [7.76 to 10.54]
  Day 1, 12 hours postdose | 5.76 [4.55 to 6.97] | 5.18 [3.93 to 6.43] | 6.93 [5.68 to 8.19]
  Day 2, 24 hours postdose | 2.32 [1.25 to 3.40] | 1.60 [0.53 to 2.67] | 2.92 [1.81 to 4.02]

4. Secondary Outcome: Change From Baseline QT Interval Using Fridericia's Formula (ΔQTcF)
Description: as for outcome 3
Time Frame: as for outcome 3
Population: as for outcome 1
Measure: Least Squares Mean (90% Confidence Interval); unit: ms
Groups:
- ALXN1840: Participants received ALXN1840 120 mg administered as 15 mg enteric-coated tablets (supratherapeutic dose). .
Arm/Group | ALXN1840 | Placebo | Moxifloxacin
Number analyzed (Participants) | 57 | 56 | 53
ms
  Day 1, 0.5 hours postdose | -2.56 [-3.52 to -1.61] | -2.36 [-3.31 to -1.40] | 2.29 [1.30 to 3.27]
  Day 1, 1 hour postdose | -0.49 [-1.49 to 0.51] | -0.19 [-1.19 to 0.82] | 9.47 [8.43 to 10.50]
  Day 1, 2 hours postdose | -0.69 [-1.81 to 0.43] | -0.76 [-1.88 to 0.35] | 10.28 [9.12 to 11.43]
  Day 1, 3 hours postdose | -1.04 [-2.11 to 0.02] | -0.41 [-1.47 to 0.66] | 10.96 [9.86 to 12.07]
  Day 1, 4 hours postdose | -1.06 [-2.29 to 0.16] | 0.02 [-1.21 to 1.25] | 10.03 [8.75 to 11.30]
  Day 1, 5 hours postdose | -0.64 [-1.89 to 0.61] | -0.55 [-1.80 to 0.71] | 9.54 [8.24 to 10.83]
  Day 1, 6 hours postdose | -6.05 [-7.52 to -4.58] | -5.35 [-6.80 to -3.89] | 4.00 [2.48 to 5.53]
  Day 1, 7 hours postdose | -7.60 [-8.92 to -6.28] | -7.85 [-9.18 to -6.52] | 2.05 [0.67 to 3.43]
  Day 1, 8 hours postdose | -7.66 [-8.86 to -6.47] | -6.73 [-7.93 to -5.53] | 1.49 [0.25 to 2.73]
  Day 1, 10 hours postdose | -4.96 [-6.34 to -3.58] | -5.73 [-7.13 to -4.33] | 1.70 [0.25 to 3.15]
  Day 1, 12 hours postdose | -5.05 [-6.61 to -3.49] | -5.10 [-6.70 to -3.50] | 0.94 [-0.68 to 2.56]
  Day 2, 24 hours postdose | 0.52 [-0.56 to 1.60] | -1.78 [-2.85 to -0.70] | 3.48 [2.37 to 4.59]

5. Secondary Outcome: Change From Baseline PR Interval (ΔPR)
Description: as for outcome 3
Time Frame: as for outcome 3
Population: as for outcome 1
Measure: Least Squares Mean (90% Confidence Interval); unit: ms
Arm/Group | ALXN1840 | Placebo | Moxifloxacin
Number analyzed (Participants) | 57 | 56 | 53
ms
  Day 1, 0.5 hours postdose | -0.13 [-1.55 to 1.29] | 1.26 [-0.16 to 2.69] | -1.33 [-2.81 to 0.14]
  Day 1, 1 hour postdose | 0.41 [-0.95 to 1.78] | 1.66 [0.29 to 3.03] | -1.37 [-2.79 to 0.04]
  Day 1, 2 hours postdose | 1.30 [0.05 to 2.56] | 1.54 [0.29 to 2.79] | -0.77 [-2.06 to 0.52]
  Day 1, 3 hours postdose | 0.46 [-0.88 to 1.79] | 1.32 [-0.01 to 2.66] | -2.66 [-4.05 to -1.28]
  Day 1, 4 hours postdose | -0.75 [-2.08 to 0.58] | -0.10 [-1.43 to 1.23] | -3.38 [-4.75 to -2.00]
  Day 1, 5 hours postdose | -1.72 [-3.14 to -0.30] | -1.12 [-2.54 to 0.31] | -4.22 [-5.70 to -2.75]
  Day 1, 6 hours postdose | -3.64 [-5.00 to -2.28] | -3.43 [-4.79 to -2.08] | -5.52 [-6.93 to -4.11]
  Day 1, 7 hours postdose | -5.76 [-7.14 to -4.38] | -4.05 [-5.44 to -2.67] | -7.16 [-8.59 to -5.72]
  Day 1, 8 hours postdose | -4.52 [-5.86 to -3.18] | -3.83 [-5.17 to -2.48] | -7.07 [-8.46 to -5.68]
  Day 1, 10 hours postdose | -3.94 [-5.57 to -2.32] | -3.34 [-4.97 to -1.69] | -6.61 [-8.30 to -4.91]
  Day 1, 12 hours postdose | -2.89 [-4.21 to -1.56] | -2.98 [-4.35 to -1.61] | -4.60 [-5.98 to -3.22]
  Day 2, 24 hours postdose | -0.13 [-1.55 to 1.29] | 0.69 [-0.73 to 2.10] | -1.68 [-3.14 to -0.21]

6. Secondary Outcome: Change From Baseline QRS Interval (ΔQRS)
Description: as for outcome 3
Time Frame: as for outcome 3
Population: as for outcome 1
Measure: Least Squares Mean (90% Confidence Interval); unit: ms
Arm/Group | ALXN1840 | Placebo | Moxifloxacin
Number analyzed (Participants) | 57 | 56 | 53
ms
  Day 1, 0.5 hours postdose | -0.01 [-0.22 to 0.21] | -0.07 [-0.29 to 0.14] | -0.08 [-0.30 to 0.14]
  Day 1, 1 hour postdose | 0.04 [-0.20 to 0.29] | -0.04 [-0.29 to 0.21] | 0.06 [-0.19 to 0.32]
  Day 1, 2 hours postdose | 0.08 [-0.20 to 0.36] | -0.09 [-0.38 to 0.19] | -0.10 [-0.39 to 0.19]
  Day 1, 3 hours postdose | 0.10 [-0.17 to 0.38] | -0.05 [-0.33 to 0.22] | -0.19 [-0.47 to 0.10]
  Day 1, 4 hours postdose | 0.14 [-0.14 to 0.43] | 0.16 [-0.13 to 0.44] | 0.01 [-0.29 to 0.30]
  Day 1, 5 hours postdose | -0.23 [-0.54 to 0.09] | -0.28 [-0.60 to 0.04] | -0.35 [-0.68 to -0.02]
  Day 1, 6 hours postdose | -1.01 [-1.31 to -0.71] | -0.73 [-1.03 to -0.44] | -1.13 [-1.44 to -0.82]
  Day 1, 7 hours postdose | -0.89 [-1.16 to -0.63] | -1.08 [-1.34 to -0.82] | -1.16 [-1.44 to -0.89]
  Day 1, 8 hours postdose | -0.66 [-0.97 to -0.35] | -0.39 [-0.69 to -0.08] | -0.48 [-0.80 to -0.16]
  Day 1, 10 hours postdose | -0.89 [-1.26 to -0.52] | -0.71 [-1.08 to -0.34] | -0.87 [-1.25 to -0.48]
  Day 1, 12 hours postdose | -0.42 [-0.74 to 0.11] | -0.30 [-0.62 to 0.02] | -0.50 [-0.83 to -0.18]
  Day 2, 24 hours postdose | -0.14 [-0.44 to 0.16] | 0.02 [-0.27 to 0.32] | -0.18 [-0.48 to 0.13]

7. Secondary Outcome: Placebo-corrected Change From Baseline Heart Rate (ΔΔHR)
Description: Twelve-lead ECGs were extracted from approximately 25-hour continuous (Holter) recordings on Day -1 of Treatment Period 1 and Days 1 and 2 in each treatment period.
  Least square mean difference and its 90% CI were calculated based on MMRM with fixed effects for period, sequence, timepoint, treatment, time-by-treatment interaction as fixed effect and baseline value and sex as covariates.
Time Frame: as for outcome 3
Population: as for outcome 1
Measure: Least Squares Mean (90% Confidence Interval); unit: bpm
Arm/Group | ALXN1840 | Moxifloxacin
Number analyzed (Participants) | 57 | 53
bpm
  Day 1, 0.5 hours postdose | -0.77 [-1.76 to 0.21] | 0.77 [-0.24 to 1.77]
  Day 1, 1 hour postdose | -0.40 [-1.52 to 0.72] | 3.50 [2.35 to 4.64]
  Day 1, 2 hours postdose | -0.31 [-1.32 to 0.69] | 1.78 [0.76 to 2.80]
  Day 1, 3 hours postdose | 1.58 [0.36 to 2.80] | 3.31 [2.07 to 4.56]
  Day 1, 4 hours postdose | 0.27 [-1.06 to 1.59] | 2.06 [0.71 to 3.42]
  Day 1, 5 hours postdose | 1.02 [-0.35 to 2.40] | 0.99 [-0.41 to 2.40]
  Day 1, 6 hours postdose | 0.13 [-1.32 to 1.58] | 0.48 [-0.99 to 1.96]
  Day 1, 7 hours postdose | 1.27 [-0.47 to 3.00] | 2.29 [0.50 to 4.07]
  Day 1, 8 hours postdose | 0.72 [-0.72 to 2.15] | 1.40 [-0.07 to 2.86]
  Day 1, 10 hours postdose | 0.27 [-1.54 to 2.09] | 1.71 [-0.15 to 3.58]
  Day 1, 12 hours postdose | 0.58 [-1.07 to 2.24] | 1.75 [0.06 to 3.45]
  Day 2, 24 hours postdose | 0.73 [-0.69 to 2.15] | 1.32 [-0.12 to 2.76]

8. Secondary Outcome: Placebo-corrected Change From Baseline PR Interval (ΔΔPR)
Description: as for outcome 3
Time Frame: as for outcome 3
Population: as for outcome 1
Measure: Least Squares Mean (90% Confidence Interval); unit: ms
Arm/Group | ALXN1840 | Moxifloxacin
Number analyzed (Participants) | 57 | 53
ms
  Day 1, 0.5 hours postdose | -1.39 [-3.29 to 0.51] | -2.60 [-4.54 to -0.66]
  Day 1, 1 hour postdose | -1.25 [-3.07 to 0.57] | -3.03 [-4.89 to -1.18]
  Day 1, 2 hours postdose | -0.24 [-1.88 to 1.41] | -2.31 [-3.98 to -0.63]
  Day 1, 3 hours postdose | -0.87 [-2.64 to 0.90] | -3.99 [-5.79 to -2.18]
  Day 1, 4 hours postdose | -0.65 [-2.41 to 1.11] | -3.28 [-5.08 to -1.48]
  Day 1, 5 hours postdose | -0.60 [-2.51 to 1.30] | -3.11 [-5.05 to -1.16]
  Day 1, 6 hours postdose | -0.21 [-2.01 to 1.60] | -2.09 [-3.93 to -0.24]
  Day 1, 7 hours postdose | -1.71 [-3.55 to 0.14] | -3.10 [-4.99 to -1.21]
  Day 1, 8 hours postdose | -0.69 [-2.48 to 1.09] | -3.24 [-5.06 to -1.42]
  Day 1, 10 hours postdose | -0.61 [-2.83 to 1.60] | -3.28 [-5.54 to -1.01]
  Day 1, 12 hours postdose | 0.09 [-1.70 to 1.89] | -1.62 [-3.46 to 0.21]
  Day 2, 24 hours postdose | -0.82 [-2.71 to 1.08] | -2.37 [-4.30 to -0.44]

9. Secondary Outcome: Placebo-corrected Change From Baseline QRS Interval (ΔΔQRS)
Description: as for outcome 7
Time Frame: as for outcome 3
Population: as for outcome 1
Measure: Least Squares Mean (90% Confidence Interval); unit: ms
Arm/Group | ALXN1840 | Moxifloxacin
Number analyzed (Participants) | 57 | 53
ms
  Day 1, 0.5 hours postdose | 0.07 [-0.21 to 0.35] | -0.01 [-0.29 to 0.28]
  Day 1, 1 hour postdose | 0.08 [-0.25 to 0.41] | 0.10 [-0.23 to 0.44]
  Day 1, 2 hours postdose | 0.17 [-0.21 to 0.56] | -0.01 [-0.40 to 0.38]
  Day 1, 3 hours postdose | 0.15 [-0.22 to 0.53] | -0.13 [-0.52 to 0.25]
  Day 1, 4 hours postdose | -0.02 [-0.40 to 0.37] | -0.15 [-0.55 to 0.24]
  Day 1, 5 hours postdose | 0.05 [-0.38 to 0.49] | -0.07 [-0.51 to 0.38]
  Day 1, 6 hours postdose | -0.27 [-0.68 to 0.13] | -0.40 [-0.81 to 0.01]
  Day 1, 7 hours postdose | 0.19 [-0.17 to 0.54] | -0.08 [-0.45 to 0.28]
  Day 1, 8 hours postdose | -0.27 [-0.69 to 0.15] | -0.10 [-0.52 to 0.33]
  Day 1, 10 hours postdose | -0.18 [-0.69 to 0.33] | -0.15 [-0.68 to 0.37]
  Day 1, 12 hours postdose | -0.12 [-0.56 to 0.31] | -0.20 [-0.65 to 0.24]
  Day 2, 24 hours postdose | -0.16 [-0.57 to 0.25] | -0.20 [-0.61 to 0.21]

10. Secondary Outcome: Number of Participants With Treatment-emergent T-wave Morphology Abnormalities and U-waves
Description: as for outcome 3
Time Frame: Day 1 (after dosing) through 24 hours postdose
Population: All participants who received at least 1 dose of study treatment with measurements at baseline as well as on-treatment with at least 1 postdose time point.
Measure: Count of Participants; unit: Participants
Arm/Group | ALXN1840 | Placebo | Moxifloxacin
Number analyzed (Participants) | 57 | 56 | 53
Participants
  At least one treatment-emergent T-wave abnormality | 0 | 0 | 1
  At least one treatment-emergent U-wave | 0 | 0 | 0

11. Secondary Outcome: ALXN1840 PK Parameter: Area Under The Concentration Versus Time Curve From Time 0 To The Last Quantifiable Concentration (AUC0-t) Of Total Molybdenum And Plasma Ultrafiltrate (PUF) Molybdenum Following a Single Oral Dose of ALXN1840
Description: Blood samples for PK analysis of total molybdenum and PUF molybdenum were collected as close as possible to nominal time after completion of the ECG extraction period.
Time Frame: Predose (0) to 96 hours post-dose
Population: All participants who received at least 1 dose of study treatment with evaluable data. It was pre-specified to collect data for only the ALXN1840 Arm for this outcome measure.
Measure: Geometric Mean (Geometric Coefficient of Variation); unit: h*ng/mL
Arm/Group | ALXN1840
Number analyzed (Participants) | 57
h*ng/mL
  Total Molybdenum | 18450 (44.5)
  Plasma Ultrafiltrate Molybdenum | 1763 (84.8)

12. Secondary Outcome: ALXN1840 PK Parameter: Maximum Observed Concentration (Cmax) Of Total Molybdenum And PUF Molybdenum Following a Single Oral Dose of ALXN1840
Description: as for outcome 11
Time Frame: Predose (0) to 96 hours post-dose
Population: as for outcome 11
Measure: Geometric Mean (Geometric Coefficient of Variation); unit: ng/mL
Arm/Group | ALXN1840
Number analyzed (Participants) | 57
ng/mL
  Total Molybdenum | 504.1 (46.8)
  Plasma Ultrafiltrate Molybdenum | 127.9 (120.5)

13. Secondary Outcome: ALXN1840 PK Parameter: Time To Maximum Observed Concentration (Tmax) Of Total Molybdenum And PUF Molybdenum Following a Single Oral Dose of ALXN1840
Description: as for outcome 11
Time Frame: Pre-dose to 96 hours post-dose
Population: as for outcome 11
Measure: Median (Full Range); unit: hours
Arm/Group | ALXN1840
Number analyzed (Participants) | 57
hours
  Total Molybdenum | 5.00 [0.52 to 8.02]
  Plasma Ultrafiltrate Molybdenum | 6.00 [3.00 to 10.00]

14. Secondary Outcome: Number of Participants With Treatment-Emergent Adverse Events (TEAEs)
Description: An adverse event (AE) was any untoward medical occurrence in a participant, temporally associated with the use of study intervention, whether or not considered related to the study intervention. TEAE was an AE that started during or after the first dose, or started prior to the first dose and increased in severity after the first dose. A related TEAE was defined as having a reasonable possibility the study intervention caused the AE as assessed by the investigator. Serious AEs were defined as any untoward medical occurrence that met at least 1 of the following serious criteria: resulted in death, was life-threatening, required in-patient hospitalization or prolongation of existing hospitalization, resulted in persistent or significant disability/incapacity, was a congenital anomaly/birth defect, other medically important serious event.
Time Frame: Day 1 (after dosing) through Day 70
Population: All participants who received at least 1 dose of study drug.
Measure: Count of Participants; unit: Participants
Arm/Group | ALXN1840 | Placebo | Moxifloxacin
Number analyzed (Participants) | 57 | 56 | 53
Participants
  Any TEAE | 9 | 3 | 6
  Any serious TEAE (SAE) | 0 | 0 | 0
  Any TEAE leading to death | 0 | 0 | 0
  Any related TEAE | 4 | 0 | 3

ADVERSE EVENTS:
Time Frame: Day 1 (after dosing) through Day 70
Groups:
- Overall: All treated participants.
Arm/Group | ALXN1840 | Placebo | Moxifloxacin | Overall
All-Cause Mortality (participants affected / at risk) | 0/57 | 0/56 | 0/53 | 0/57
Serious Adverse Events (participants affected / at risk) | 0/57 | 0/56 | 0/53 | 0/57
Other Adverse Events (participants affected / at risk) | 9/57 | 3/56 | 6/53 | 16/57
OTHER ADVERSE EVENTS; cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | ALXN1840 (N=57) | Placebo (N=56) | Moxifloxacin (N=53) | Overall (N=57)
Tinnitus (Ear and labyrinth disorders) | 1 (1) | 0 (0) | 1 (1) | 2 (2)
Abdominal discomfort (Gastrointestinal disorders) | 1 (1) | 0 (0) | 0 (0) | 1 (1)
Abdominal pain (Gastrointestinal disorders) | 1 (1) | 0 (0) | 0 (0) | 1 (1)
Dyspepsia (Gastrointestinal disorders) | 0 (0) | 1 (1) | 0 (0) | 1 (1)
Eructation (Gastrointestinal disorders) | 0 (0) | 1 (1) | 0 (0) | 1 (1)
Gastrointestinal sounds abnormal (Gastrointestinal disorders) | 0 (0) | 0 (0) | 1 (1) | 1 (1)
Nausea (Gastrointestinal disorders) | 1 (1) | 0 (0) | 3 (3) | 4 (4)
Proctalgia (Gastrointestinal disorders) | 1 (1) | 0 (0) | 0 (0) | 1 (1)
Fatigue (General disorders) | 0 (0) | 0 (0) | 1 (1) | 1 (1)
Feeling cold (General disorders) | 1 (1) | 0 (0) | 0 (0) | 1 (1)
Feeling of body temperature change (General disorders) | 0 (0) | 0 (0) | 1 (1) | 1 (1)
Hordeolum (Infections and infestations) | 1 (1) | 0 (0) | 0 (0) | 1 (1)
Pustule (Infections and infestations) | 0 (0) | 0 (0) | 1 (1) | 1 (1)
Urinary tract infection (Infections and infestations) | 0 (0) | 1 (1) | 0 (0) | 1 (1)
Chemical burns of eye (Injury, poisoning and procedural complications) | 0 (0) | 0 (0) | 1 (1) | 1 (1)
SARS-CoV-2 test positive (Investigations) | 1 (1) | 0 (0) | 0 (0) | 1 (1)
Musculoskeletal discomfort (Musculoskeletal and connective tissue disorders) | 0 (0) | 0 (0) | 1 (1) | 1 (1)
Pain in extremity (Musculoskeletal and connective tissue disorders) | 0 (0) | 1 (1) | 0 (0) | 1 (1)
Dizziness (Nervous system disorders) | 1 (1) | 0 (0) | 2 (2) | 3 (3)
Headache (Nervous system disorders) | 2 (2) | 0 (0) | 0 (0) | 2 (2)
Oropharyngeal pain (Respiratory, thoracic and mediastinal disorders) | 1 (1) | 0 (0) | 0 (0) | 1 (1)
Rhinitis allergic (Respiratory, thoracic and mediastinal disorders) | 1 (1) | 0 (0) | 0 (0) | 1 (1)
Dermatitis contact (Skin and subcutaneous tissue disorders) | 0 (0) | 0 (0) | 1 (1) | 1 (1)

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: Yes

DOCUMENTS (2):
  • Study Protocol (2020-09-01): https://cdn.clinicaltrials.gov/large-docs/16/NCT04560816/Prot_000.pdf
  • Statistical Analysis Plan (2020-09-03): https://cdn.clinicaltrials.gov/large-docs/16/NCT04560816/SAP_001.pdf